CLINICAL TRIAL: NCT06397625
Title: Short- and Medium-term Efficacy of Treatment With Peripheral Nerve Stimulation of the Pudendal Nerve in Patients With Erectile Dysfunction: a Randomized Clinical Trial
Brief Title: Treatment With Peripheral Nerve Stimulation of the Pudendal Nerve in Patients With Erectile Dysfunction
Acronym: NEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NEEP
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction; Electric Stimulation; Pudendal Nerve
Keywords: Erectile Dysfunction; Percutaneous Electrical Neurostimulation; Pudendal Nerve
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (Placebo) (Placebo Comparator): Group I (Control), will be operated with the same procedure but without electric current, and using "placebo needles" of the same size (Streitberger Placebo-Needle ® , Asiamed, Pullach, Germany), which will not pierce the surface of the patient's skin, but will cause a prick sensation. This process will be developed by resting the needle on the skin of the patient's perineum and pushing the handle of the needle until it touches the surface of the skin, producing in the patient the impression of penetration, although this is not the case.
  Interventions: Other: Percutaneous electrical neurostimulation (Placebo)
- Group (20 Hertz) (Experimental): Group II will undergo continuous stimulation at a frequency of 20 Hertz, a pulse width of 200 μs and for a total of 20 minutes. The intensity will be set at the maximum tolerated by the patient.
  Interventions: Other: Percutaneous electrical neurostimulation
- Group 3 (50 Hertz) (Experimental): Group III, will be intervened with continuous stimulation at a frequency of 50 Hz,a pulse width of 200 μs (18) and for a total of 20 minutes. The intensity will be set at the maximum tolerable threshold. In case the patient does not tolerate the treatment, due to increased fatigue, the 50 hertz will be alternated with the 20 hertz in bursts.
  Interventions: Other: Percutaneous electrical neurostimulation

INTERVENTIONS:
Other: Percutaneous electrical neurostimulation (Placebo) — Group I (Control), will be operated with the same procedure but without electric current, and using "placebo needles" of the same size (Streitberger Placebo-Needle ® , Asiamed, Pullach, Germany)
  Arms: Group (Placebo)
Other: Percutaneous electrical neurostimulation — The Group II and III electrostimulation procedure is called peripheral nerve stimulation and is known as an echo-guided peripheral nerve stimulation technique using a blunt, dry needle (active electrode). The intervention will be performed on the pudendal nerve, in an area where there is no risk of perforating any vascular-nerve bundle. The invasive technique will be performed by a physiotherapist expert in musculoskeletal and peripheral nervous system ultrasound and specialized in invasive techniques, with two years of experience in the sector. The needle will be introduced through the anterior (perineum).
  Arms: Group (20 Hertz); Group 3 (50 Hertz)

SUMMARY:
Erectile dysfunction is known as any alteration that produces a modification in the erectile response, whether of organic, psychogenic or relational cause. In this case the pudendal nerve is addressed, since it has its origin in the sacral plexus, deriving from the S2, S3 and S4 nerve branches. Its fibers have different innervation, being the pudendal nerve a mixed nerve, and estimating that it has 30% of autonomic innervation, and 70% of somatic innervation (50% sensory and 20% motor). Peripheral percutaneous nerve stimulation (proposed treatment) is performed with a needle to stimulate the peripheral nerves in such a way as to stimulate most of the area of the structure, stimulating sensory and motor nerve endings of the deeper tissues.

DETAILED DESCRIPTION:
The study corresponds to an experimental, prospective, multicenter, randomized, prospective clinical trial. According to the Granmo program, it has been calculated to recruit 72 subjects with erectile dysfunction, recruited from different leading urology and andrology centers such as Clínica LYX (Instituto de Urología de Madrid). Patients will voluntarily accept to be part of the study, and will be able to ask the principal investigator any questions they may have at any time. The intervention will be performed at the LYX Clinic (Urology Institute).

ELIGIBILITY:
Inclusion Criteria:

* Men
* Ages 18-60 years old
* Primarily organic cause diagnosed by Doppler:

Peak-systolic velocities (PSV). Tele-diastolic velocity (DTV). Resistance Index (IR)

* Initial IIEF-EF questionnaire scores: 1-25 points (mild, moderate or severe erectile dysfunction).
* Active sex life (more than 4 attempts per month).

Exclusion Criteria:

* Pelvic surgeries
* History of Peyronie's disease
* Penile surgeries, except circumcision or frenuloplasty
* Priapism
* Pelvic radiation
* Women

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF-EF) | 4 months
  It is an index that assesses erectile function in a purely subjective way. It is the most widely recognized and used, and consists of six questions in which the frequency and firmness of erection, penetration capacity, capacity and frequency of maintenance and confidence in erection are evaluated. According to the questionnaire, dysfunction is classified as: no ED (26-30 points), mild (22-25 points), mild to moderate (17-21 points), moderate (11-16 points) and very strong (6-10 points). A score equal to or greater than 4 points will be considered a significant change. Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention.
Erection Hardness Scale (EHS) | 4 months
  significant changes will be considered to be those men who improved by more than 3 points what in the initial phase was below a score of 2 points. The questionnaire score depends on the rating of erection hardness according to the following parameters: 0 (penis does not enlarge); 1 (penis is larger, but not hard); 2 (penis is hard but not hard enough for penetration); 3 (penis is hard enough to penetrate, but not completely hard); and 4 (penis is completely hard and rigid). Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention.
Intravaginal Latency Time (IELT) | 4 months
  Time to ejaculation is considered and should be between 3 and 6 minutes. A duration of less than one minute is considered premature ejaculation, and a duration between one minute and one and a half minutes is considered probable premature ejaculation. Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention.
Premature Ejaculation Diagnostic Tool (PEDT) | 4 months
  Helps identify patients who may be suffering from premature ejaculation. Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention.
Quality of Life Scale | 4 months
  It is used to know in a subjective way, the patient's opinion regarding his/her quality of life, according to 4 main aspects: physical, psychological, social and environmental health. Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention. The scale is measured by 26 items, divided into 4 dimensions. Each dimension is independent. The higher the score, the higher the patient's quality of life.
Self-Esteem And Relationship Questionnaire (Sear) | 4 months
  It is a questionnaire used for research and/or clinical practice on self-esteem, in this case for patients with erectile dysfunction. Measurement pre-, one week after the intervention, one month after the intervention and 3 months after the intervention. The scale is measured from 0 to 100 points, with 0 being the worst score and 100 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Navas Mosqueda, Principal Investigator — Camilo Jose Cela Univerity
Locations (1):
- LYX Instituto de Urología, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rislanu A, Auwal H, Musa D, Auwal A. Comparative Effectiveness of Electrical Stimulation and Aerobic Exercise in the Management of Erectile Dysfunction: A Randomized Clinical Trial. Ethiop J Health Sci. 2020 Nov;30(6):961-970. doi: 10.4314/ejhs.v30i6.14. PMID 33883841
- [Background] Carboni C, Fornari A, Bragante KC, Averbeck MA, Vianna da Rosa P, Mea Plentz RD. An initial study on the effect of functional electrical stimulation in erectile dysfunction: a randomized controlled trial. Int J Impot Res. 2018 Jun;30(3):97-101. doi: 10.1038/s41443-018-0024-8. Epub 2018 May 22. PMID 29785045
- [Background] Yafi FA, Jenkins L, Albersen M, Corona G, Isidori AM, Goldfarb S, Maggi M, Nelson CJ, Parish S, Salonia A, Tan R, Mulhall JP, Hellstrom WJ. Erectile dysfunction. Nat Rev Dis Primers. 2016 Feb 4;2:16003. doi: 10.1038/nrdp.2016.3. PMID 27188339